CLINICAL TRIAL: NCT00751673
Title: A Prospective, Multicentre Study Evaluating the Clinical Performance of the T.E.S.S Anatomic and Reverse Shoulder Prostheses
Brief Title: TESS Shoulder Arthroplasty Data Collection
Status: Terminated | Type: Observational
Why Stopped: No more data collected.
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet France SARL (Industry)
Responsible Party: Sponsor
Other Study IDs: BMETEU.CR.EU74
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TESS prosthesis: Consecutive series of patients with a TESS prosthesis.

SUMMARY:
This observational study intends to collect efficacy and safety data on TESS shoulder system

DETAILED DESCRIPTION:
The T.E.S.S.® shoulder system has been developed to provide a complete solution for all the indications for Shoulder Arthroplasty, Arthritis, Rotator Cuff Arthropathy, Proximal Humeral Fracture, minimising bone resection and restoring the natural anatomy of the patient.

ELIGIBILITY:
Inclusion Criteria:

* A pre-operative level of pain and function the same as for conventional joint replacement
* A likelihood of obtaining relief of pain and improved function
* Full skeletal maturity
* Ability to follow instructions
* Good general health for age
* Willing to return for follow-up evaluations

Exclusion Criteria:

* Glenohumeral joint infection, osteomyelitis
* Neuro-muscular complications
* Inability to co-operate with and complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of patients received TESS prostheses
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2006-01; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change in Constant Murley Score | 6 months, 1 year, 2 year, 3 year, 4 year, 5 year, 7 year and 10 year
  Improvement in this score will be collected at every follow-up visit.This is a 100-point score, containing 8 questions. Higher score indicate a better outcome.
Change in Oxford Score | 6 months, 1 year, 2 year, 3 year, 4 year, 5 year, 7 year and 10 year
  Improvement in this score will be collected at every follow-up visit.This is a 60-point score, containing 12 questions. Higher score indicate a better outcome.

SECONDARY OUTCOMES:
Complications | Any time
  General and shoulder specific complicatons are collected any time.
Patient Satisfaction | 6 months, 1 year, 2 year, 3 year, 4 year, 5 year, 7 year and 10 year
  Binary question.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BEGUIN, MD, Principal Investigator — Clinique Mutualiste (Saint Etienne)
Locations (13):
- De Dreef Van Zonnebos 13, Schilde, Belgium
- France (12):
  - Clinique Générale, Annecy
  - Institut Calot, Berck
  - Polyclinique Jean Villar, Bruges
  - Clinique St Joseph, Chambéry
  - Centre Hospitalier Général, Dax
  - Clinique Chirurgicale Orthopédique A.D.R., Maxéville
  - Clinique St Jean, Montpellier
  - IRCOS, Paris
  - Clinique St Martin, Pessac
  - Clinique Mutualiste, Saint-Etienne
  - Polyclinique de l'Atlantique, Saint-Herblain
  - Institut A. Tzanck, Saint-Laurent-du-Var